CLINICAL TRIAL: NCT02507843
Title: Vitamin D as an Adjunctive Treatment in Patients With Non-Cystic Fibrosis Bronchiectasis: a Double-blind Randomised Controlled Trial
Brief Title: Vitamin D as an Adjunctive Treatment in Patients With Non-Cystic Fibrosis Bronchiectasis
Acronym: VIDB
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, MD, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20150511
Record Dates: First submitted 2015-07-22; First posted 2015-07-24 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Bronchiectasis
Keywords: Vitamin D
MeSH Terms: conditions — Bronchiectasis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D group (Active Comparator): Cholecalciferol will be administered by monthly oral intake. During a prospective follow-up period of one year, the patients will get the normal care with some additional tests for the study.
  Interventions: Drug: Cholecalciferol
- Placebo group (Placebo Comparator): Placebo will be administered by monthly oral intake. During a prospective follow-up period of one year, the patients will get the normal care with some additional tests for the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — Oral Cholecalciferol(100000 IU) will be administered in Vitamin D group monthly for 6 months.
  Other Names: Vitamin D3
  Arms: Vitamin D group
Drug: Placebo — Placebo will be administered in placebo group monthly for 6 months.
  Other Names: Migliol Placebo Oil
  Arms: Placebo group

SUMMARY:
This study evaluates vitamin D as an adjunctive treatment in patients with non-Cystic Fibrosis bronchiectasis, which are combined with vitamin D deficiency. Half of participants will receive vitamin D supplementation, while the other half will receive placebo.

DETAILED DESCRIPTION:
To define the therapeutic effect of Vitamin D in the treatment of non-Cystic Fibrosis bronchiectasis by means of a prospective randomized placebo-controlled double blind study with a follow-up of at least one year. To explore whether correction of Vitamin D deficiency by the oral supplementation of Vitamin D triggers the vitamin D receptors-mediated cathelicidin pathway and increases local or systemic concentrations of the natural antimicrobial polypeptide cathelicidin with enhanced eradication of bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-Cystic fibrosis bronchiectasis by High Resolution CT
* Age 18 years or older
* Vitamin D deficiency [25(OH)D<20 ng/mL]
* Informed consent

Exclusion Criteria:

* Current active allergic bronchopulmonary or tuberculosis
* Diagnosis of any of the following: sarcoidosis, hyperparathyroidism, nephrolithiasis, pulmonary silicosis, Human Immunodeficiency Virus infection, liver failure, renal failure or malignancy
* Taking benzothiadiazine derivative, cardiac glycoside, carbamazepine, phenobarbital, phenytoin or primidone
* Taking dietary supplement or topical preparation containing vitamin D up to 2 months before first dose
* Treatment with any investigational medical product or device up to 4 months before first dose
* Breastfeeding, pregnant or planning a pregnancy
* Baseline corrected serum calcium > 2.65 mmol/L
* Baseline serum creatinine > 125 micromol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Time to first acute exacerbation | one year

SECONDARY OUTCOMES:
total number of exacerbations per group | one year
percentage of patients with one or more exacerbations per year | one year
severity of diseases | one year
  FACED（FEV1% predicted, age, chronic colonization by Pseudomonas aeruginosa， radiological extent of the disease， and dyspnea） score
using of antibiotics | one year
  types of antibiotics used during exacerbations
quality of life | one year
  the Quality of Life-Bronchiectasis (QOL-B) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: JinFu Xu, Principal Investigator — Shanghai Pulmonary Hospital , Tongji University
Locations (1):
- Shanghai Pulmonary Hospital , Tongji University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Chalmers JD, McHugh BJ, Docherty C, Govan JR, Hill AT. Vitamin-D deficiency is associated with chronic bacterial colonisation and disease severity in bronchiectasis. Thorax. 2013 Jan;68(1):39-47. doi: 10.1136/thoraxjnl-2012-202125. Epub 2012 Oct 16. PMID 23076388
- [Result] Bartley J, Garrett J, Grant CC, Camargo CA Jr. Could vitamin d have a potential anti-inflammatory and anti-infective role in bronchiectasis? Curr Infect Dis Rep. 2013 Apr;15(2):148-57. doi: 10.1007/s11908-013-0321-9. PMID 23371406
- [Result] Martinez-Garcia MA, de Gracia J, Vendrell Relat M, Giron RM, Maiz Carro L, de la Rosa Carrillo D, Olveira C. Multidimensional approach to non-cystic fibrosis bronchiectasis: the FACED score. Eur Respir J. 2014 May;43(5):1357-67. doi: 10.1183/09031936.00026313. Epub 2013 Nov 14. PMID 24232697